CLINICAL TRIAL: NCT00192829
Title: Hypercoagulable Parameters as Predictors of Thrombotic Events and Prognosis in Patients With Advanced Non-Small Cell Lung Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Other Study IDs: Thrombosis and cancer.CTIL
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2007-04-11 (Estimated); Status verified 2007-03

CONDITIONS: Non-Small Cell Lung Carcinoma; Venous Thromboembolism
Keywords: Lung cancer; Thrombosis; Hypercoagulable
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Venous Thromboembolism; Lung Neoplasms; Thrombosis; Thrombophilia

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Procedure: Blood sample withdrawal

SUMMARY:
The association between cancer and thrombosis is well known and the occurrence of thrombotic complications is commonly associated with poor prognosis. The aim os this study is to determine the possible value of hypercoagulable parameters as prognostic parameters in advanced non-small cell lung carcinoma (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of NSCLC.
* normal serum bilirubin
* informed concent to participate in the study

Exclusion Criteria:

* anticoagulant therapy
* infectious disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100
Dates: Start 2005-06

CONTACTS AND LOCATIONS:
Overall Officials: Galit Sarig, Ph.D, Principal Investigator — Rambam Health Care Campus
Locations (2):
- Israel (2):
  - Hematology Laboratory, Haifa
  - Oncology Institution, Rambam Health Campus, Haifa

REFERENCES:
- [Background] Haim N, Lanir N, Hoffman R, Haim A, Tsalik M, Brenner B. Acquired activated protein C resistance is common in cancer patients and is associated with venous thromboembolism. Am J Med. 2001 Feb 1;110(2):91-6. doi: 10.1016/s0002-9343(00)00691-4. PMID 11165549
- [Background] Blom JW, Osanto S, Rosendaal FR. The risk of a venous thrombotic event in lung cancer patients: higher risk for adenocarcinoma than squamous cell carcinoma. J Thromb Haemost. 2004 Oct;2(10):1760-5. doi: 10.1111/j.1538-7836.2004.00928.x. PMID 15456487
- [Background] Ferrigno D, Buccheri G, Ricca I. Prognostic significance of blood coagulation tests in lung cancer. Eur Respir J. 2001 Apr;17(4):667-73. doi: 10.1183/09031936.01.17406670. PMID 11401062